CLINICAL TRIAL: NCT05232357
Title: In Vivo Evaluation of Tumor Neurogenesis in Gastrointestinal Diseases by Topical Submucosal Chromoendoscopy
Brief Title: Endoscopic Vital Nerve Staining in Gastrointestinal Diseases
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Endoscopic nerve staining
Record Dates: First submitted 2022-01-05; First posted 2022-02-09 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-02

CONDITIONS: Gastrointestinal Neoplasms; Abnormality of Enteric Nervous System Morphology
Keywords: Endoscopy; Gastrointestinal Neoplasms; Enteric Nervous System; Gastric nervous system; nerve staining; Methylene blue
MeSH Terms: conditions — Gastrointestinal Neoplasms | interventions — sodium thiosulfate; Methylene Blue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Endoscopic nerve staining (Experimental): Methylene blue (MB) solution was used as nerve staining agent. Routine endoscopic submucosal injection of MB solution for mucosal nerve staining was used to identify and evaluate the neural architecture and special morphology of normal gastrointestinal mucosa, adenoma and malignant lesions.
  Interventions: Drug: Sodium thiosulfate and Methylene blue solution

INTERVENTIONS:
Drug: Sodium thiosulfate and Methylene blue solution — Take a methylene blue injection (2ml:20mg), add 18ml distilled water and mix well. Add NaS2O3.5H2O800mg to the methylene blue solution 10ml, add 4 drops of dilute hydrochloric acid, heat the water bath until the dark blue fades, the solution is milky and turbid, adjust the PH to about 3.5. Put the prepared solution into a glass bottle with a rubber stopper, which is wrapped in tin foil, sealed and protected from light, and stored in a refrigerator at-20 ℃. It can be used after high-pressure sterilization before operation. Sodium thiosulfate-Methylene blue (DMB) staining solution was used as nerve staining agent. During gastroenteroscopy, DMB staining solution was locally sprayed on the surface of gastrointestinal lesion mucosa or injected into the lesion mucosa.
  Other Names: NaS2O3.5H2O and Methylene blue injection (2ml:20mg)

SUMMARY:
In this study, methylene blue (MB) was used as vital nerve staining agent. During gastroenteroscopy, mucosal nerve staining was achieved by endoscopic submucosal injection of MB solution. To observe the staining of nerve fibers, neurons and glial cells in mucosa and submucosa, as well as the morphological changes, density differences and function of mucosal nerve tissues in different gastrointestinal lesions, in order to explore the role of endoscopic vital nerve staining in the diagnosis of gastrointestinal lesions.

DETAILED DESCRIPTION:
This study is a prospective experimental study. The baseline data of the patients were recorded objectively: sex, age, vital signs, body weight, some laboratory examination results (blood routine, liver function, blood coagulation function and electrolytes, etc.) and related medical history (comorbidities, treatment history and life history). Mucosal nerve staining was achieved by endoscopic submucosal injection of methylene blue (MB) solution. The following features were identified and then compared between normal, adenoma and neoplastic mucosa on magnifying endoscopy images in vivo: nerve morphology (straight or irregular), nerve diameter, branching patterns and nerve density. Immunohistochemistry was used to further confirm the presence and to study the morphology of neural structures (PGP9.5 and GFAP staining) and neural attribute (VIP, nNOS, TH, ChAT and SOM staining) on tumor, adenoma and normal mucosal sections.The aim of this study was to explore the role of MB based topical submucosal chromoendoscopy in the identification of neural architecture and special morphology in normal gastrointestinal mucosa, adenomas and malignant lesions during routine endoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis or suspected diagnosis of one of the following common gastrointestinal diseases: chronic non-atrophic gastritis, chronic atrophic gastritis, gastric polyps, gastric early cancer, advanced gastric cancer; colonic polyps, colonic Melanosis, early colon cancer, advanced colon cancer
2. Written informed consent

Exclusion Criteria:

1. Those who are allergic to nerve dye components (such as methylene blue, etc.)
2. Complicated with cardiovascular and cerebrovascular diseases, or severely impaired liver, kidney and hematopoietic system.
3. Psychopath
4. There are hemorrhagic diseases
5. Platelet count < 50 × 10 ^ 9 / L
6. Those who are allergic to body mass are
7. Unable to tolerate or cooperate with endoscopy
8. Patients with serious complications, such as severe infection, gastrointestinal bleeding, obstruction and perforation, etc.
9. Pregnant or lactating women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-05-01 (Estimated); Study Completion 2022-05-15 (Estimated)

PRIMARY OUTCOMES:
Morphological characteristics of mucosal nerves in different gastrointestinal lesions | Immediately after operation
  Mucosal nerve staining was achieved by endoscopic submucosal injection of MB solution. The following features were identified and then compared between normal, adenoma and neoplastic mucosa on magnifying endoscopy images in vivo: nerve morphology (straight or irregular), nerve diameter, branching patterns and nerve density.
Expression levels of PGP9.5, GFAP, VIP, nNOS, TH, ChAT and SOM of different gastrointestinal lesions | 1 to 3 days after operation
  Immunohistochemistry was used to further confirm the presence and to study the morphology of neural structures (PGP9.5 and GFAP staining) and neural attribute (VIP, nNOS, TH, ChAT and SOM staining) on tumor, adenoma and normal mucosal sections.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Liu, MD, Principal Investigator — Beijing 302 Hospital
Locations (1):
- The First Medical Center of Chinese PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No